CLINICAL TRIAL: NCT02689648
Title: Long Term Follow up on Functional Gastrointestinal Disorder (FGID)
Acronym: LUFT
Status: Active, not recruiting | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Staffan Berglund, MD, PhD, Umeå University
Other Study IDs: LUFT2016
Record Dates: First submitted 2016-02-08; First posted 2016-02-24 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Functional Gastrointestinal Disorder
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Long term prognosis and risk factors in functional gastrointestinal disorder (FGID) is largely unknown. The investigators plan to retrospectively analyse a cohort of children who were referred to the Pediatric Clinic due to abdominal pain with the aims to learn more about symptoms and effects of investigations performed. Furthermore, the investigators plan to contact the cases for a follow up using a validated questionnaire and analyse the long term prognosis and risk factors for prolonged severe symptoms.

DETAILED DESCRIPTION:
Long term prognosis and risk factors in functional gastrointestinal disorder (FGID) is largely unknown. The investigators plan to retrospectively analyse a cohort of children who during the years 2010-2015 were referred to the Pediatric Clinic of Umeå University Hospital due to abdominal pain. The aims are to explore and descriptively describe the symptoms and effects of investigations performed. Furthermore, the investigators plan to contact the cases five years after the first contact for a follow up using a validated questionnaire of the ROME-III-criteria and analyse the long term prognosis and risk factors for prolonged severe symptoms.

ELIGIBILITY:
At time of first visit the children had:

1. At least 2 months of abdominal pain
2. Age 3-18 years
3. No organic gastrointestinal diseases
4. No neuromuscular disease

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children between 3 and 18 years of age that were refereed to the Pediatric Clinic of Västerbotten county council during the years 2009-2015.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-02; Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of patients that fulfill the ROME-III criteria for FGID | 5 years after fist visit +/- 1 year
  Measured by the validated ROME-III questionnaire

SECONDARY OUTCOMES:
ICD 10-diagnosis following the primary investigation | 12 months after first visit
Current ICD 10-diagnosis | 5 years after fist visit +/- 1 year
Number (n) of visits for the primary investigations | 0-12 months after first visit

CONTACTS AND LOCATIONS:
Overall Officials: Staffan K Berglund, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Department of Clinical Sciences, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No